CLINICAL TRIAL: NCT03206801
Title: A Randomized Controlled Trial of Urine CXCL10 Chemokine Monitoring Post-renal Transplant
Brief Title: Urine CXCL10 Monitoring Trial in Kidney Transplant
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian National Transplant Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: B2017:076; 364003 (Other Grant/Funding Number: Canadian Institutes of Health Research); TMCT-04 (Other: Transplant Manitoba)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Complications; Rejection of Renal Transplant
Keywords: Urine biomarker; CXCL10 chemokine; Post-transplant monitoring; Protocol biopsy

STUDY DESIGN:
Intervention Model Description: This is a Phase II-III multi-center prospective randomized controlled clinical trial of incident adult renal transplant patients. Patients with elevated urine CXCL10 will be randomized 1:1 to the intervention and control arms, stratified by center (~ 420 enrolled to urine CXCL10 screening for n=250 randomized participants).
Who Masked: Outcomes Assessor
Masking Description: The assessor of the primary outcome will be masked. As the intervention involves a study biopsy, based on an elevated urine CXCL10, it is not possible to blind the participant, care provider or investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants with high urine CXCL10 randomized to the Intervention Arm will undergo a kidney transplant biopsy to check for rejection. Biopsy-proven subclinical rejection will be treated per study protocol.
  Interventions: Procedure: Kidney transplant biopsy
- Control (No Intervention): Participants with high urine CXCL10 randomized to the Control Arm will continue routine post-transplant surveillance with serum creatinine and proteinuria; serial urine samples will continue to be collected and analyzed (blinded), but not used to direct care.

INTERVENTIONS:
Procedure: Kidney transplant biopsy — Elevated urine CXCL10 will trigger a study biopsy in patients randomized to the intervention arm. Subclinical rejection will be treated per protocol.
  Other Names: Protocol biopsy
  Arms: Intervention

SUMMARY:
This is a Phase II-III multi-center prospective randomized controlled clinical trial of incident adult renal transplant patients.

The primary objective of this study is to determine if the early treatment of rejection, as detected by urinary CXCL10, will improve renal allograft outcomes.

DETAILED DESCRIPTION:
This is a Phase II-III multi-center prospective randomized controlled clinical trial of incident adult renal transplant patients. Patients will be screened for eligibility (n≈485) and n≈420 will be enrolled and undergo post-transplant surveillance with urinary CXCL10. Two hundred and fifty patients deemed at high risk for rejection based on a confirmed elevated urine CXCL10 will undergo 1:1 randomization to the intervention and control arms, stratified by center. The total study duration is approximately 5 years; and there two main phases - screening and intervention.

All eligible, enrolled patients will undergo the Screening Phase (n≈420). Routine urine CXCL10 screening will be done from 2 weeks - 9 months post-transplant. We have previously shown that urine CXCL10 is elevated in ischemia-reperfusion injury, so screening will commence at 2 weeks (+/- 4 days) to exclude this as a potential confounding factor (60).

If patient develops a confirmed elevated urine CXCL10 level and is considered high risk for rejection, they will proceed to Randomization in the Intervention Phase, which can occur anytime between 2 weeks - 9 months post-transplant. Participants in the Intervention Arm will undergo renal biopsy to check for rejection. Biopsy-proven subclinical rejection will be treated per study protocol. Participants in the Control Arm will continue routine post-transplant surveillance with serum creatinine and proteinuria; serial urine samples will continue to be collected and analyzed (blinded), but not used to direct care. All randomized participants will undergo a 12-month study exit visit with protocol biopsy to determine primary, secondary and long-term outcomes.

Enrolled patients with persistently low urine CXCL10 and low risk of rejection from 2 weeks - 9 months post-transplant will be considered Off-Study (not randomized). They will undergo a 12-month study exit visit (+/- 7 days) to determine secondary and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to understand and provide written informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. All ethnic and gender groups will have equal access to the study
4. Incident adult (age ≥18) renal transplant patients with a living or deceased donor kidney transplant
5. Confirmed elevated urine CXCL10:Cr without a urinary tract infection or gross hematuria.

Exclusion Criteria:

1. Primary non-function
2. Blood group (ABO) incompatible
3. Pre-transplant donor specific antibody (DSA) positive (MFI>1000 OR positive flow crossmatch)
4. Human leukocyte (HLA) 0 HLA antigen D-related (DR) + 0 major HLA class 2 (DQ) mismatch
5. Presence of other transplanted organ or co-transplanted organ
6. Medical contraindication to biopsy or rejection treatment
7. Followed outside of investigational center
8. Participation in other interventional trials within 4-weeks post-transplant or anytime post-transplant till study end at 12-months
9. Intention to not use a maintenance immunosuppression regimen consisting of calcineurin inhibitor (CNI) and anti-proliferative agents
10. Any condition that, in the opinion of the investigator, would pose risk to the subject's safe participation, or interfere with their ability to comply with the study requirements, or may impact the quality of interpretation of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Death-censored graft loss | 2 weeks-12 months post-transplant
  Return to dialysis or re-transplant
Clinical indication biopsy-proven acute rejection | 2 weeks-12 months post-transplant
  Clinical rejection, Banff criteria
De novo donor specific antibody development | 2 weeks-12 months post-transplant
  De novo human leukocyte antibody (HLA) antibodies, donor specific
Subclinical tubulitis | 12-month study exit biopsy
  Subclinical rejection, Banff criteria
Interstitial fibrosis and inflammation (IFTA + i) | 12-month study exit biopsy
  IFTA + i, defined by Mayo criteria

SECONDARY OUTCOMES:
Renal allograft function | 6, 12, 24 and 60 months post-transplant
  Change in eGFR (slope, ∆) and graft function (eGFR) (absolute, mL/min)
Microvascular inflammation | 12-month study exit biopsy
  Banff ptc, g, c4d, cg
Development IFTA from implantation to 12-months | 12-month study exit biopsy
  Banff ∆ ci, ct, cv
Days from transplantation to clinical-biopsy proven rejection | 2 weeks-12 months post-transplant
  Time to biopsy proven rejection
Albuminuria >300mg/day | 6, 12, 24 and 60 months post-transplant
  Urine albumin: Cr ratio
Cost-effectiveness of urine CXCL10 monitoring strategy | 2 weeks-12 months post-transplant
  Costs of urine CXCL10 screening
Quality of life | 6 and 12 months post-transplant
  EuroQOL (EQ-5DL)
Urine CXCL10 kinetics | 2 weeks-12 months post-transplant
  Change in urine CXCL10 levels in response to rejection therapy

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ho, MD, Principal Investigator — University of Manitoba
Locations (9):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Transplant Manitoba Adult Kidney Program, Winnipeg, Manitoba
  - Western University, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - University Health Network, University of Toronto, Toronto, Ontario
  - Centre de recherche du CHUM (CRCHUM), Montreal, Quebec
  - McGill, Montreal, Quebec
  - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho J, Rush DN, Karpinski M, Storsley L, Gibson IW, Bestland J, Gao A, Stefura W, HayGlass KT, Nickerson PW. Validation of urinary CXCL10 as a marker of borderline, subclinical, and clinical tubulitis. Transplantation. 2011 Oct 27;92(8):878-82. doi: 10.1097/TP.0b013e31822d4de1. PMID 21876477
- [Background] Hirt-Minkowski P, Amico P, Ho J, Gao A, Bestland J, Hopfer H, Steiger J, Dickenmann M, Burkhalter F, Rush D, Nickerson P, Schaub S. Detection of clinical and subclinical tubulo-interstitial inflammation by the urinary CXCL10 chemokine in a real-life setting. Am J Transplant. 2012 Jul;12(7):1811-23. doi: 10.1111/j.1600-6143.2012.03999.x. Epub 2012 Mar 5. PMID 22390571
- [Background] Blydt-Hansen TD, Gibson IW, Gao A, Dufault B, Ho J. Elevated urinary CXCL10-to-creatinine ratio is associated with subclinical and clinical rejection in pediatric renal transplantation. Transplantation. 2015 Apr;99(4):797-804. doi: 10.1097/TP.0000000000000419. PMID 25222013
- [Background] Hirt-Minkowski P, Ho J, Gao A, Amico P, Koller MT, Hopfer H, Rush DN, Nickerson PW, Schaub S. Prediction of Long-term Renal Allograft Outcome By Early Urinary CXCL10 Chemokine Levels. Transplant Direct. 2015 Sep 24;1(8):e31. doi: 10.1097/TXD.0000000000000537. eCollection 2015 Sep. PMID 27500231
- [Background] Hirt-Minkowski P, Rush DN, Gao A, Hopfer H, Wiebe C, Nickerson PW, Schaub S, Ho J. Six-Month Urinary CCL2 and CXCL10 Levels Predict Long-term Renal Allograft Outcome. Transplantation. 2016 Sep;100(9):1988-96. doi: 10.1097/TP.0000000000001304. PMID 27548845
- [Background] Ho J, Sharma A, Mandal R, Wishart DS, Wiebe C, Storsley L, Karpinski M, Gibson IW, Nickerson PW, Rush DN. Detecting Renal Allograft Inflammation Using Quantitative Urine Metabolomics and CXCL10. Transplant Direct. 2016 May 19;2(6):e78. doi: 10.1097/TXD.0000000000000589. eCollection 2016 Jun. PMID 27500268
- [Background] Ho J, Rush DN, Krokhin O, Antonovici M, Gao A, Bestland J, Wiebe C, Hiebert B, Rigatto C, Gibson IW, Wilkins JA, Nickerson PW. Elevated Urinary Matrix Metalloproteinase-7 Detects Underlying Renal Allograft Inflammation and Injury. Transplantation. 2016 Mar;100(3):648-54. doi: 10.1097/TP.0000000000000867. PMID 26906940
- [Background] Hricik DE, Nickerson P, Formica RN, Poggio ED, Rush D, Newell KA, Goebel J, Gibson IW, Fairchild RL, Riggs M, Spain K, Ikle D, Bridges ND, Heeger PS; CTOT-01 consortium. Multicenter validation of urinary CXCL9 as a risk-stratifying biomarker for kidney transplant injury. Am J Transplant. 2013 Oct;13(10):2634-44. doi: 10.1111/ajt.12426. Epub 2013 Aug 22. PMID 23968332
- [Background] Rabant M, Amrouche L, Lebreton X, Aulagnon F, Benon A, Sauvaget V, Bonifay R, Morin L, Scemla A, Delville M, Martinez F, Timsit MO, Duong Van Huyen JP, Legendre C, Terzi F, Anglicheau D. Urinary C-X-C Motif Chemokine 10 Independently Improves the Noninvasive Diagnosis of Antibody-Mediated Kidney Allograft Rejection. J Am Soc Nephrol. 2015 Nov;26(11):2840-51. doi: 10.1681/ASN.2014080797. Epub 2015 May 6. PMID 25948873
- [Derived] Ho J, Sharma A, Kroeker K, Carroll R, De Serres S, Gibson IW, Hirt-Minkowski P, Jevnikar A, Kim SJ, Knoll G, Rush DN, Wiebe C, Nickerson P. Multicentre randomised controlled trial protocol of urine CXCL10 monitoring strategy in kidney transplant recipients. BMJ Open. 2019 Apr 11;9(4):e024908. doi: 10.1136/bmjopen-2018-024908. PMID 30975673